CLINICAL TRIAL: NCT00206050
Title: A Randomized, Open-Label, Comparative, Two-Treatment, Crossover Study of the 24-Hour Intragastric pH Profile After 5 Days of Once Daily Oral Administration of Either Esomeprazole 40 mg or Pantoprazole 40 mg Following Once Daily Infusion of Intravenous Pantoprazole 40 mg for 5 Days in Healthy Volunteer Subjects
Brief Title: Study of Intragastric pH Profile After 5 Days Pantoprazole 40 mg iv Followed by Oral Esomeprazole 40 mg po or Oral Pantoprazole 40 mg po
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D9612L00066
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole; Pantoprazole

INTERVENTIONS:
Drug: Esomeprazole
Drug: pantoprazole

SUMMARY:
This Phase IV study is intended to compare intragastric acid suppression of oral esomeprazole (NEXIUM ® Delayed-Release Capsules) with that of oral pantoprazole (PROTONIX ® Delayed Release Tablets ), in subjects who continue to require acid-suppressive therapy following a course of intravenous (iv) pantoprazole (PROTONIX ® I.V. for Injection).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Males and females aged 18 to 70 years, inclusive.
* Male or non-pregnant, nonlactating female healthy volunteer subjects. Females must be post-menopausal, surgically sterilized, or using a medically acceptable form of birth control, as determined by the investigator. Women of childbearing potential must agree to continue using an acceptable form of birth control throughout the conduct of the study.

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the investigational site)
* Previous enrollment or randomization of treatment in the present study.
* Received an experimental drug or used an experimental device within 28 days preceeding the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The percent time of intragastric pH>4.0 on oral dosing Day 5 during the 24-hour intragastric pH monitoring period.

SECONDARY OUTCOMES:
The percent time of intragastric pH>4.0 on oral dosing Day 1 and the mean hourly cumulative IGA during the 24-hour intragastric pH monitoring periods (on oral dosing Days 1 and 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Oklahoma City, Oklahoma, United States